CLINICAL TRIAL: NCT04741529
Title: Massed and Spaced Healthy Minds Program App Dosage Study
Brief Title: Massed and Spaced HMP App Dosage Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2020-1454; A171600 (Other: UW Madison); EDUC/COUNSELING PSYCH (Other: UW Madison); Protocol Approval 1/11/2021 (Other: UW Madison)
Record Dates: First submitted 2021-01-29; First posted 2021-02-05 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Depression, Anxiety; Psychological Distress; Loneliness
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Massed condition (Experimental): Participant will be asked to use the HMP app for 20 minutes per day in one 20-minute meditation session.
  Interventions: Behavioral: Healthy Minds Program app
- Spaced condition (Experimental): Participant will be asked to use the HMP app for 20 minutes per day in two 10-minute meditation sessions.
  Interventions: Behavioral: Healthy Minds Program app

INTERVENTIONS:
Behavioral: Healthy Minds Program app — The HMP app was developed by Healthy Minds Innovations at the UW Center for Healthy Minds, and is based on the work of Drs. Richard Davidson and Cortland Dahl. HMP is designed to promote and protect psychological well-being through sustainable skills training. The program is grounded in constituents of psychological well-being identified in empirical literature. HMP provides core content, with instruction administered through a curriculum of high-quality guided practices. HMP is based on research on eudaimonic well-being (e.g., environmental mastery, purpose) and brain-based skills that underlie these qualities (e.g., regulation of attention, mental flexibility). HMP has >100 guided audio practices that address 4 constituents of well-being: awareness, connection, insight, and purpose.
  Participants in this study will receive 2 weeks of training in the Connection module of HMP.

SUMMARY:
This study is a randomized controlled trial (RCT) of 2 weeks of the Healthy Minds Program (HMP) app Connection module in undergraduate students of a large, midwestern state university in the United States during the spring of 2021.

Participants will be recruited via email and/or flyers and will first complete an online screen. Eligible participants will complete baseline measures prior to attending an introductory session via web conferencing. During this session, participants will be randomly assigned to condition. Participants in both conditions will be asked to use the HMP app for 20 minutes per either, either split over two 10-minute session (Spaced condition) or in one 20-minute session (Massed condition). Participants will complete daily survey measures during the study and post-test measures after 2 weeks of intervention.

This study is primarily designed to assess feasibility and acceptability of 2 weeks of Connection training and assignment to dosage condition. Study team will investigate self-reported informal practice on the daily diary measure, measures of psychological distress (composite of depression, anxiety) and loneliness.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Undergraduate at UW-Madison
* Access to a smartphone or device capable of downloading HMP app
* PROMIS Depression or PROMIS Anxiety ≥55

Exclusion Criteria:

* Meditation retreat experience
* Regular meditation practice (i.e., weekly practice for >1 year OR daily practice within previous 6 months)
* Previous practice under the instruction of a meditation teacher, other than in the context of an introductory course
* PROMIS Depression ≥70

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2021-05-18 (Actual); Study Completion 2021-05-18 (Actual)

PRIMARY OUTCOMES:
Percentage of participants who completed the study | 2 weeks
Number of meditation sessions per day using the HMP app | 2 weeks
Number of minutes of meditation practice using the HMP app | 2 weeks
System Usability Scale score | 2 weeks
  System usability scale is (SUS) is a 10-item Likert scale questionnaire that provides information on the ease of use (or lack thereof) of websites, software, hardware, mobile devices, and other technological applications. Higher SUS score correlates to better usability of an app, total score range = 0 to 100

SECONDARY OUTCOMES:
Change in the PROMIS (Patient-Reported Outcomes Measurement Information System) Depression score | Baseline and 2 weeks
  Psychological distress computed as composite of 4-item PROMIS Depression measures. Scores range from 4 to 20 with higher scores representing worse symptoms.
Change in the PROMIS Anxiety score | Baseline and 2 weeks
  Psychological distress computed as composite of 4-item PROMIS Anxiety measures. Scores range from 4 to 20 with higher scores representing worse symptoms.
Change in NIH Toolbox Loneliness score | Baseline and 2 weeks
  NIH toolbox loneliness measures the perceptions that one is alone, lonely, or socially isolated from others. It is a 5-item scale. Total score range = 5 to 25, lower score is better
Change in Self-Compassion Short Form score | Baseline and 2 weeks
  This 12-item measure assesses participant's self-compassion ability, total score range = 12 to 60, higher scores correlate to more self-compassion.
Change in Fear of Missing Out scale score | Baseline and 2 weeks
  Fear of missing out is a 10 item scale. Total score range = 10 to 50, lower score is better
Change in Acceptance and Action Questionnaire - II score | Baseline and 2 weeks
  Acceptance and Action Questionnaire- II measures psychological flexibility Experiential avoidance, total score range = 7 to 49. Higher total scores mean less flexibility, while lower total scores mean more flexibility. Lower score is better.
Single item loneliness score | Up to 2 weeks
  "How lonely did you feel today?", range = 1 to 7, lower score is better
Highest loading PROMIS Depression and PROMIS Anxiety items score | Up to 2 weeks
  Composite of highest loading PROMIS items modified to reference "today," z-transformed to have mean of 0 and standard deviation of 1, lower score is better.
Single item informal meditation practice | Up to 2 weeks
  Single item informal meditation practice measure, "As you reflect on today, to what extent did you apply these practices?" Scores range from 0 to 100. A higher score is better.
Digital Working Alliance Inventory score | 2 weeks
  The Digital Working Alliance Inventory measures the therapeutic relationship between participant and HMP app. Total score range = 6 to 42, higher score is better.

CONTACTS AND LOCATIONS:
Overall Officials: Simon B Goldberg, PhD, Principal Investigator — UW-Madison
Locations (1):
- University of Wisconsin - Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be de-identified and listed in public data registries (i.e., osf) based on the publication of preregistered study hypotheses on a manuscript by manuscript basis.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data may be shared following analysis and publication or upon request.

REFERENCES:
- [Derived] Riordan KM, Simonsson O, Frye C, Vack NJ, Sachs J, Fitch D, Goldman RI, Chiang ES, Dahl CJ, Davidson RJ, Goldberg SB. How often should I meditate? A randomized trial examining the role of meditation frequency when total amount of meditation is held constant. J Couns Psychol. 2024 Mar;71(2):104-114. doi: 10.1037/cou0000725. PMID 38376930